CLINICAL TRIAL: NCT06638450
Title: Dense Cranial Electroacupuncture Stimulation Plus Body Acupuncture for Adolescents With Psychological Distress: a Randomized Controlled Trial With Observations on Salivary Oxytocin and Cortisol Changes
Brief Title: Clinical Trial for Acupuncture in Adolescents With Psychological Distress and Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Group of Hospitals (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 24-333
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Psychological Distress; Insomnia
Keywords: Psychological distress; Insomnia; Acupuncture; Adolescent
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCEAS+BA group (Experimental): Subjects assigned to Dense Cranial Electroacupuncture Stimulation plus Body Acupuncture (DCEAS+BA) group will receive DCEAS+BA treatment, twice weekly for 8 weeks, in addition to their current interventions and medications as usual.
  Interventions: Procedure: Dense Cranial Electroacupuncture Stimulation plus Body Acupuncture (DCEAS+BA)
- MAS group (Sham Comparator): Subjects assigned to Minimal Acupuncture Stimulation (MAS) group will receive MAS treatment, twice weekly for 8 weeks, in addition to their current interventions and medications as usual.
  Interventions: Procedure: Minimal Acupuncture Stimulation (MAS)

INTERVENTIONS:
Procedure: Dense Cranial Electroacupuncture Stimulation plus Body Acupuncture (DCEAS+BA) — DCEAS+BA will be conducted for 2 sessions per week for 8 weeks.
  For DCEAS, 6 pairs of acupoints are used: Baihui (GV20) and Yintang (EX-HN3), left Sishencong (EX-HN1) and Toulinqi (GB15), right Sishencong (EX-HN1) and Toulinqi (GB15), bilateral Shuaigu (GB8), bilateral Taiyang (EX-HN5), and bilateral Touwei (ST8). For body acupuncture, the following acupoints are used: Shenmen (HT7). Neiguan (PC6), Zhongwan (CV12), Guanyuan (CV4), Zusanli (ST36), Sanyinjiao (SP6), and Taichong (LV3).
  Disposable acupuncture needles (0.25 mm in diameter and 25-40 mm in length) are inserted at a depth of 10-30 mm perpendicularly or obliquely into acupoints. Manual manipulation is conducted to evoke a needling sensation. After that, electrical stimulation is delivered on DCEAS, with continuous waves at 2 Hz through an electrical acupuncture stimulation instrument (Hwarto, SDZ-II). The stimulation lasts 30 minutes.
  Arms: DCEAS+BA group
Procedure: Minimal Acupuncture Stimulation (MAS) — MAS will be conducted for 2 sessions per week for 8 weeks.
  The following 6 acupoints are used: bilateral Tongtian (BL07), bilateral Shousanli (LI10) and bilateral Fuyang (BL59).
  Disposable acupuncture needles (0.25 mm in diameter and 25-40 mm in length) are inserted at a depth of 10-30 mm perpendicularly or obliquely into acupoints. After that, electrical stimulation is performed on bilateral Tongtian (BL07), with continuous waves at 2 Hz through an electrical acupuncture stimulation instrument (Hwarto, SDZ-II). The stimulation lasts 30 minutes.
  Arms: MAS group

SUMMARY:
This is an assessor-blinded, randomized, MAS-controlled trial. A total of 148 adolescents aged 15-22 years experiencing mild to moderate anxiety or depressive symptoms will be recruited. They will be randomly assigned to DCEAS+BA (n = 74) and MAS (n = 74) for 2 sessions per week for 8 weeks, followed by a 4-week post-treatment observation period. A post-intervention visit will be held at week 12. The primary outcome will be assessed using the Chinese version of the Beck Anxiety Inventory (BAI-C). The secondary outcomes include the Beck Depression Inventory II (C-BDI-II) for depression, the Zung Self-Rating Anxiety Scale (SAS) and the Zung Self-Rating Depression Scale (SDS) as additional assessments for anxiety and depression, the Pittsburgh Sleep Quality Index (PSQI) for sleep quality, and the World Health Organization Quality of Life-Brief (WHOQOL-BREF) (HK version) for the general quality of life. Assessment will be carried out every 4 weeks till week 12, while saliva will be collected at baseline and at the end of the 8 weeks. Salivary oxytocin and cortisol will be analyzed. A generalized linear mixed-effect model will be applied to compare treatment outcomes over time in the two groups and linear regression will be conducted to examine intercorrelations among clinical improvement and changes in biomarker levels. Subgroup analysis will be conducted to identify specific effects of DCEAS+BA.

DETAILED DESCRIPTION:
Psychological distress refers to a state of emotional suffering characterized by symptom(s) including anxiety, depression, and stress, and is often accompanied by somatic symptoms such as insomnia, headache, and lack of energy. As subclinical symptoms or clinical diagnoses, anxiety and depression are often core symptoms in psychological distress. They are highly comorbid and are often accompanied by physical and sleep problems. Psychological distress is particularly prevalent in adolescents and can be a precursor or features of various psychiatric disorders. One epidemiological study conducted in Hong Kong local university students has revealed that approximately 70% of students complained of some degree of depression and 54% of anxiety; nearly 9% had moderately severe to severe depressive symptoms and 6% had severe anxiety. Two most recent large-scale surveys respectively conducted in Hong Kong and China further revealed about 17% of children and youths probably had a mental problem. This has become more severe during and post COVID-19 pandemic. However, psychiatric disorders of youths are often underdiagnosed and vastly undertreated, because the condition of most young patients is mild and they may fear drugs' side effects which sometimes are a greater risk than the disease itself. This has led to particularly low acceptability for medication interventions in adolescents. The development of novel non-pharmacological treatment strategies for youth is therefore greatly desired.

A large body of evidence well confirms the benefits and effectiveness of acupuncture in the treatment of depression, anxiety, and various related disorders. Recently, we further developed a novel acupuncture mode called 'dense cranial electroacupuncture stimulation plus body acupuncture (DCEAS+BA)', where "dense" represents the use of many acupoints mainly located on the forehead. DCEAS is a novel nerve stimulation that is established based on neuroanatomical rationales, i.e., electrical stimulation is conducted on many forehead acupoints that are innervated by the first branch of the trigeminal nerve. We have demonstrated the effectiveness of DCEAS in the treatment of major depression, post-stroke cognitive impairment, insomnia, obsessive-compulsive disorder (OCD), and chemotherapy-induced cognitive impairment. Previous studies also have revealed that transcutaneous trigeminal nerve stimulation is eﬀective in reducing depression, anxiety, attention-deﬁcit/hyperactivity disorder (ADHD) and epilepsy. Compared to adults, adolescents are more sensitive to peripheral nerve stimulation, producing robust neuromodulatory effects. These have led to the hypothesis that DCEAS+BA may have particular effects in alleviating adolescents' psychological distress.

Saliva collection is highly acceptable for children and adolescents. Salivary oxytocin and cortisol are the two most compelling biomarkers for screenings, diagnoses, and predicting treatment outcomes in children and adolescents with psychiatric disorders. Children and adolescents with social disorder and emotional distress had significantly lower levels of salivary oxytocin and higher cortisol levels. Electroacupuncture and acupuncture suppressed salivary cortisol levels while anxiety symptoms were alleviated. The oxytocin system plays an important role in the therapeutic mechanisms of acupuncture in the treatment of pain disorders and autism. These studies suggest that salivary oxytocin and cortisol could serve as valid biomarkers for predicting the treatment outcomes of acupuncture.

Over the past years, we have completed a series of clinical trials evaluating the efficacy of acupuncture, with particular DCEAS+BA in patients with cognitive impairment, depression, and insomnia. However, our previous studies of DCEAS mainly focused on the general population with psychiatric disorders and aged subjects with stroke, and only estimated clinical efficacy, but did not explore associations with specific biomarker profiles. In particular, it is not yet validated in young subjects with psychological distress.

There have been several lines of evidence suggesting that younger subjects with psychiatric disorders could achieve earlier responses and may be more efficacious for nerve and brain stimulation compared to older adults. There also exists an age difference in the analgesic effects of electroacupuncture between adult and juvenile rats. On the other hand, meta-analysis and recent trials suggested that acupuncture and electroacupuncture may have more benefits in treating anxiety disorders and insomnia, and produce comparable efficacy in improving anxiety disorders as compared to anxiolytics. This has led to the anticipation that youths with psychological distress could achieve better outcomes on DCEAS+BA compared to other subpopulations. Therefore, we further propose this trial to examine the efficacy of DCEAS+BA and its associations with salivary oxytocin and cortisol in adolescents with psychological distress. As youths with psychiatric disorders are vastly undertreated, are often reluctant and even decline to take the medications due to fear of the drugs' side effects, the validation of the efficacy of DCEAS+BA provides an effective and acceptable option for this special subpopulation. The exploration of the associations with biomarkers will help us gain more insights into the mechanisms of DCEAS.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for this study if they:

1. are experiencing anxiety as evidenced by a BAI-C score of at least 8 (no symptoms = 0-7; mild = 8-15; moderate = 16-25; severe = 26-63), and/or a C-BDI-II score of at least 14 (no symptoms = 0-13, mild = 14-19; moderate = 20-28; severe = 29-63);
2. have symptoms that have persistent for more than 3 months;
3. are able to provide informed consent for participation, and complete treatments and questionnaires as scheduled; and
4. have no suicidal ideation, as evidenced by "no" answers or a score of <3 for all questionnaires of the Columbia-Suicide Severity Rating Scale (C-SSRS).

Exclusion Criteria:

Subjects will be excluded if they:

1. have unstable systemic medical conditions that may limit their participation in the study, for example, severe liver, cardiovascular, or kidney impairment; gastrointestinal or endocrine dysfunction; malignancy; autoimmune disease; acute infectious disease; or any conditions with unstable vital signs or require intensive hospitalization;
2. have bipolar or psychotic disorder (e.g. schizophrenia);
3. have a history of brain injury or surgery;
4. have alcohol abuse or substance abuse;
5. are pregnant or in lactation, or intend to conceive;
6. have heart pacemaker or other metal devices implanted in the body;
7. have concurrent or use of drug treatment for anxiety/depression in the previous 6 months;
8. have treatment with acupuncture or brain stimulation in the previous 6 months;
9. have a history of epilepsy;
10. have a condition of bleeding tendency, or coagulopathy, or currently receiving anti-coagulant treatment; or
11. involved in other interventional clinical studies in the last 3 months or any relevant condition potentially interfering with study evaluation.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in the Beck Anxiety Inventory score | Baseline, Week 4, Week 8, Week 12
  Beck Anxiety Inventory (BAI-C) is used to measure the severity of anxiety and its overall score ranges from 0 to 63. A higher score indicates greater severity. Assessments will be conducted at baseline, week 4, week 8 and week 12 (post-intervention visit).

SECONDARY OUTCOMES:
Change in the Beck Depression Inventory-II score | Baseline, Week 4, Week 8, Week 12
  Beck Depression Inventory-II (C-BDI-II) is used to measure the severity of depression and its overall score ranges from 0 to 63. A higher score indicates greater severity. Assessments will be conducted at baseline, week 4, week 8 and week 12 (post-intervention visit).
Change in the Zung Self-Rating Anxiety Scale score | Baseline, Week 4, Week 8, Week 12
  Zung Self-Rating Anxiety Scale (SAS) is used to measure the severity of anxiety and its overall score ranges from 25 to 100. A higher score indicates greater severity. Assessments will be conducted at baseline, week 4, week 8 and week 12 (post-intervention visit).
Change in the Zung Self-Rating Depression Scale score | Baseline, Week 4, Week 8, Week 12
  Zung Self-Rating Depression Scale (SDS) is used to measure the severity of depression and its overall score ranges from 25 to 100. A higher score indicates greater severity. Assessments will be conducted at baseline, week 4, week 8 and week 12 (post-intervention visit).
Change in the Pittsburgh Sleep Quality Index score | Baseline, Week 4, Week 8, Week 12
  Pittsburgh Sleep Quality Index (PSQI) is used to assess sleep quality and its overall score ranges from 0 to 21. A higher score indicates more acute sleep disturbances. Assessments will be conducted at baseline, week 4, week 8 and week 12 (post-intervention visit).
Change in the World Health Organization Quality of Life-Brief (HK version) score | Baseline, Week 4, Week 8, Week 12
  World Health Organization Quality of Life-Brief (WHOQOL-BREF) (HK version) is used to assess quality of life, with four quality of life domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items). Each individual item is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. A higher score indicates better quality of life. Assessments will be conducted at baseline, week 4, week 8 and week 12 (post-intervention visit).
Salivary oxytocin level | Baseline and Week 8
  Salivary samples will be collected at baseline and 8-week respectively. On collection day, 2 salivary samples will be collected in 08:00-09:00 and 20:00-21:00, respectively, to meet the cortisol circadian rhythm with peak time at 08:30 and the lowest level at 20:00-22:00. Volume of each sample collected is 3-4 ml and the detailed procedure is described in assay kit. Oxytocin and cortisol concentrations will be analyzed using enzyme-linked immunosorbent assay (ELISA) kits.
Salivary cortisol level | Baseline and Week 8
  Salivary samples will be collected at baseline and 8-week respectively. On collection day, 2 salivary samples will be collected in 08:00-09:00 and 20:00-21:00, respectively, to meet the cortisol circadian rhythm with peak time at 08:30 and the lowest level at 20:00-22:00. Volume of each sample collected is 3-4 ml and the detailed procedure is described in assay kit. Oxytocin and cortisol concentrations will be analyzed using enzyme-linked immunosorbent assay (ELISA) kits.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin Zhang, MMed, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen CJ, Chen YC, Ho CS, Lee YC. Effects of preferred music therapy on peer attachment, depression, and salivary cortisol among early adolescents in Taiwan. J Adv Nurs. 2019 Sep;75(9):1911-1921. doi: 10.1111/jan.13975. Epub 2019 Mar 13. PMID 30746740
- [Background] Briel A, Veber B, Dureuil B. [Selenium deficiency favors the appearance of heart failure after multiple injury]. Ann Fr Anesth Reanim. 1997;16(7):911-2. doi: 10.1016/s0750-7658(97)89841-3. French. PMID 9750622
- [Background] Cook IA, Abrams M, Leuchter AF. Trigeminal Nerve Stimulation for Comorbid Posttraumatic Stress Disorder and Major Depressive Disorder. Neuromodulation. 2016 Apr;19(3):299-305. doi: 10.1111/ner.12399. Epub 2016 Jan 28. PMID 26818103
- [Background] Cotovio G, Boes AD, Press DZ, Oliveira-Maia AJ, Pascual-Leone A. In Older Adults the Antidepressant Effect of Repetitive Transcranial Magnetic Stimulation Is Similar but Occurs Later Than in Younger Adults. Front Aging Neurosci. 2022 Jul 19;14:919734. doi: 10.3389/fnagi.2022.919734. eCollection 2022. PMID 35928992
- [Background] DeGiorgio CM, Soss J, Cook IA, Markovic D, Gornbein J, Murray D, Oviedo S, Gordon S, Corralle-Leyva G, Kealey CP, Heck CN. Randomized controlled trial of trigeminal nerve stimulation for drug-resistant epilepsy. Neurology. 2013 Feb 26;80(9):786-91. doi: 10.1212/WNL.0b013e318285c11a. Epub 2013 Jan 30. PMID 23365066
- [Background] Enck P, Klosterhalfen S, Zipfel S. Acupuncture, psyche and the placebo response. Auton Neurosci. 2010 Oct 28;157(1-2):68-73. doi: 10.1016/j.autneu.2010.03.005. Epub 2010 Apr 1. PMID 20359961
- [Background] Gordon I, Zagoory-Sharon O, Schneiderman I, Leckman JF, Weller A, Feldman R. Oxytocin and cortisol in romantically unattached young adults: associations with bonding and psychological distress. Psychophysiology. 2008 May;45(3):349-52. doi: 10.1111/j.1469-8986.2008.00649.x. Epub 2008 Feb 4. PMID 18266803
- [Background] Han JS. Acupuncture: neuropeptide release produced by electrical stimulation of different frequencies. Trends Neurosci. 2003 Jan;26(1):17-22. doi: 10.1016/s0166-2236(02)00006-1. No abstract available. PMID 12495858
- [Background] Ho CY, Lee A. Cultivating a Healthy Living Environment for Adolescents in the Post-COVID Era in Hong Kong: Exploring Youth Health Needs. Int J Environ Res Public Health. 2022 Jun 9;19(12):7072. doi: 10.3390/ijerph19127072. PMID 35742326
- [Background] Huang W, Taylor A, Howie J, Robinson N. Is the diurnal profile of salivary cortisol concentration a useful marker for measuring reported stress in acupuncture research? A randomized controlled pilot study. J Altern Complement Med. 2012 Mar;18(3):242-50. doi: 10.1089/acm.2010.0325. Epub 2012 Mar 2. PMID 22385023
- [Background] Kohlhoff J, Cibralic S, Hawes DJ, Eapen V. Oxytocin receptor gene (OXTR) polymorphisms and social, emotional and behavioral functioning in children and adolescents: A systematic narrative review. Neurosci Biobehav Rev. 2022 Apr;135:104573. doi: 10.1016/j.neubiorev.2022.104573. Epub 2022 Feb 9. PMID 35149102
- [Background] Lebowitz ER, Leckman JF, Feldman R, Zagoory-Sharon O, McDonald N, Silverman WK. Salivary oxytocin in clinically anxious youth: Associations with separation anxiety and family accommodation. Psychoneuroendocrinology. 2016 Mar;65:35-43. doi: 10.1016/j.psyneuen.2015.12.007. Epub 2015 Dec 14. PMID 26716876
- [Background] Li F, Cui Y, Li Y, Guo L, Ke X, Liu J, Luo X, Zheng Y, Leckman JF. Prevalence of mental disorders in school children and adolescents in China: diagnostic data from detailed clinical assessments of 17,524 individuals. J Child Psychol Psychiatry. 2022 Jan;63(1):34-46. doi: 10.1111/jcpp.13445. Epub 2021 May 21. PMID 34019305
- [Background] Li L, Lok GKI, Mei SL, Cui XL, An FR, Li L, Cheung T, Ungvari GS, Xiang YT. Prevalence of depression and its relationship with quality of life among university students in Macau, Hong Kong and mainland China. Sci Rep. 2020 Sep 25;10(1):15798. doi: 10.1038/s41598-020-72458-w. PMID 32978428
- [Background] Notkins AL, Prabhakar BS. Monoclonal autoantibodies that react with multiple organs. Basis for reactivity. Ann N Y Acad Sci. 1986;475:123-34. doi: 10.1111/j.1749-6632.1986.tb20862.x. PMID 3024548
- [Background] Man SC, Hung BH, Ng RM, Yu XC, Cheung H, Fung MP, Li LS, Leung KP, Leung KP, Tsang KW, Ziea E, Wong VT, Zhang ZJ. A pilot controlled trial of a combination of dense cranial electroacupuncture stimulation and body acupuncture for post-stroke depression. BMC Complement Altern Med. 2014 Jul 19;14:255. doi: 10.1186/1472-6882-14-255. PMID 25038733
- [Background] McGough JJ, Sturm A, Cowen J, Tung K, Salgari GC, Leuchter AF, Cook IA, Sugar CA, Loo SK. Double-Blind, Sham-Controlled, Pilot Study of Trigeminal Nerve Stimulation for Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2019 Apr;58(4):403-411.e3. doi: 10.1016/j.jaac.2018.11.013. Epub 2019 Jan 28. PMID 30768393
- [Background] Schrader LM, Cook IA, Miller PR, Maremont ER, DeGiorgio CM. Trigeminal nerve stimulation in major depressive disorder: first proof of concept in an open pilot trial. Epilepsy Behav. 2011 Nov;22(3):475-8. doi: 10.1016/j.yebeh.2011.06.026. Epub 2011 Aug 4. PMID 21820361
- [Background] Yamashita H, Zeredo JLL, Toda K. Age Differences in Naloxone Reversibility of Electroacupuncture on the Jaw Opening Reflex in Rats. J Acupunct Meridian Stud. 2021 Aug 31;14(4):167-172. doi: 10.51507/j.jams.2021.14.4.167. PMID 35770559
- [Background] Yang J, Yang Y, Chen JM, Liu WY, Wang CH, Lin BC. Effect of oxytocin on acupuncture analgesia in the rat. Neuropeptides. 2007 Oct;41(5):285-92. doi: 10.1016/j.npep.2007.05.004. Epub 2007 Jul 30. PMID 17664006
- [Background] Yang XY, Yang NB, Huang FF, Ren S, Li ZJ. Effectiveness of acupuncture on anxiety disorder: a systematic review and meta-analysis of randomised controlled trials. Ann Gen Psychiatry. 2021 Jan 30;20(1):9. doi: 10.1186/s12991-021-00327-5. PMID 33516258
- [Background] Yeung WF, Chung KF, Poon MM, Ho FY, Zhang SP, Zhang ZJ, Ziea ET, Wong VT. Acupressure, reflexology, and auricular acupressure for insomnia: a systematic review of randomized controlled trials. Sleep Med. 2012 Sep;13(8):971-84. doi: 10.1016/j.sleep.2012.06.003. Epub 2012 Jul 25. PMID 22841034
- [Background] Yeung WF, Yu BY, Yuen JW, Ho JYS, Chung KF, Zhang ZJ, Mak DSY, Suen LK, Ho LM. Semi-Individualized Acupuncture for Insomnia Disorder and Oxidative Stress: A Randomized, Double-Blind, Sham-Controlled Trial. Nat Sci Sleep. 2021 Jul 21;13:1195-1207. doi: 10.2147/NSS.S318874. eCollection 2021. PMID 34321944
- [Background] Zhang J, Qin Z, So TH, Chang TY, Yang S, Chen H, Yeung WF, Chung KF, Chan PY, Huang Y, Xu S, Chiang CY, Lao L, Zhang ZJ. Acupuncture for chemotherapy-associated insomnia in breast cancer patients: an assessor-participant blinded, randomized, sham-controlled trial. Breast Cancer Res. 2023 Apr 26;25(1):49. doi: 10.1186/s13058-023-01645-0. PMID 37101228
- [Background] Zhang J, Qin Z, So TH, Chen H, Lam WL, Yam LL, Yan Chan P, Lao L, Zhang ZJ. Electroacupuncture Plus Auricular Acupressure for Chemotherapy-Associated Insomnia in Breast Cancer Patients: A Pilot Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211019103. doi: 10.1177/15347354211019103. PMID 34036813
- [Background] Zhang ZJ, Man SC, Yam LL, Yiu CY, Leung RC, Qin ZS, Chan KS, Lee VHF, Kwong A, Yeung WF, So WKW, Ho LM, Dong YY. Electroacupuncture trigeminal nerve stimulation plus body acupuncture for chemotherapy-induced cognitive impairment in breast cancer patients: An assessor-participant blinded, randomized controlled trial. Brain Behav Immun. 2020 Aug;88:88-96. doi: 10.1016/j.bbi.2020.04.035. Epub 2020 Apr 16. PMID 32305573
- [Background] Zhang ZJ, Ng R, Man SC, Li TY, Wong W, Tan QR, Wong HK, Chung KF, Wong MT, Tsang WK, Yip KC, Ziea E, Wong VT. Dense cranial electroacupuncture stimulation for major depressive disorder--a single-blind, randomized, controlled study. PLoS One. 2012;7(1):e29651. doi: 10.1371/journal.pone.0029651. Epub 2012 Jan 6. PMID 22238631
- [Background] Zhang ZJ, Wang XM, McAlonan GM. Neural acupuncture unit: a new concept for interpreting effects and mechanisms of acupuncture. Evid Based Complement Alternat Med. 2012;2012:429412. doi: 10.1155/2012/429412. Epub 2012 Mar 8. PMID 22474503
- [Background] Zhang ZJ, Wang XY, Tan QR, Jin GX, Yao SM. Electroacupuncture for refractory obsessive-compulsive disorder: a pilot waitlist-controlled trial. J Nerv Ment Dis. 2009 Aug;197(8):619-22. doi: 10.1097/NMD.0b013e3181b05fd1. PMID 19684500
- [Background] Zhang ZJ, Zhang SY, Yang XJ, Qin ZS, Xu FQ, Jin GX, Hou XB, Liu Y, Cai JF, Xiao HB, Wong YK, Zheng Y, Shi L, Zhang JN, Zhao YY, Xiao X, Zhang LL, Jiao Y, Wang Y, He JK, Chen GB, Rong PJ. Transcutaneous electrical cranial-auricular acupoint stimulation versus escitalopram for mild-to-moderate depression: An assessor-blinded, randomized, non-inferiority trial. Psychiatry Clin Neurosci. 2023 Mar;77(3):168-177. doi: 10.1111/pcn.13512. Epub 2022 Dec 21. PMID 36445151
- [Background] Zhang ZJ, Zhao H, Jin GX, Man SC, Wang YS, Wang Y, Wang HR, Li MH, Yam LL, Qin ZS, Yu KT, Wu J, Ng FB, Ziea TE, Rong PJ. Assessor- and participant-blinded, randomized controlled trial of dense cranial electroacupuncture stimulation plus body acupuncture for neuropsychiatric sequelae of stroke. Psychiatry Clin Neurosci. 2020 Mar;74(3):183-190. doi: 10.1111/pcn.12959. Epub 2019 Dec 20. PMID 31747095